CLINICAL TRIAL: NCT00046540
Title: Liposome Encapsulated SN38 (LE-SN38) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE-SN38-101
Record Dates: First submitted 2002-09-30; First posted 2002-10-02 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasms
Keywords: Liposome-Encapsulated SN38; Irinotecan; CPT-11; Malignant Tumors
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: Liposome-encapsulated SN38

SUMMARY:
Liposome Encapsulated SN38 (LE-SN38) is an oncology drug product consisting of the active metabolite of irinotecan (CPT-11), a known anticancer drug, encapsulated in a liposome. Formulation of a relatively insoluble compound (SN38) and improvement in drug delivery (pharmacodynamic profile) may be obtained with liposomal formulations. An improved safety and efficacy profile, compared with the pro-drug CPT-11, may be possible. This rationale is supported by the results from animal toxicity studies in both the mouse and dog.

LE-SN38 will be infused intravenously every 3 weeks to assess safety and tolerability of study drug until there is disease progression or toxicity requiring early treatment discontinuation. Disease status will be assessed after every second cycle of treatment. In the event of disease progression, study treatment will be discontinued, all end-of-treatment study evaluations will be performed and further treatment options will be reviewed.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of LE-SN38.

II. Determine the plasma pharmacokinetics of SN38 following IV administration of LE-SN38.

III. Observe any anti-tumor effects of LE-SN38.

PROTOCOL OUTLINE:

This is an open-label study in patients with advanced solid tumors who have failed conventional therapy.

LE-SN38 will be administered IV over 90 minutes. At least three patients will be studied at each dose level and at least three patients will complete one 21-day course before any patient is enrolled at the next dose level. Study drug administration will continue on an every 21-day schedule in the absence of progressive disease or unacceptable toxicity. A subsequent course of treatment may be administered at least 21 days after receiving a prior dose of LE-SN38 when study criteria are met.

Cohorts of 3 patients per dose level will be studied. This will be expanded to 6 if a DLT occurs, followed by a total of 6 patients at a possible MTD.

Disease status will be assessed after every second cycle. In the event of disease progression, study treatment will be discontinued and all end of treatment study evaluations will be performed.

PROJECTED ACCRUAL: Up to 40 patients will be enrolled.

ELIGIBILITY:
Disease Characteristics:

* Advanced (local and/or metastatic) histologically documented solid tumors
* Disease not considered responsive to available conventional modalities or treatments
* No life prolonging therapy or therapy with a greater potential for patient benefit is available

Prior/Concurrent Therapy:

* No treatment with cytotoxic or biologic agents within 3 weeks prior to study entry (6 weeks for radiotherapy, mitomycin and nitrosoureas)
* At least 2 weeks since any prior surgery or hematopoietic growth factor therapy
* Chronic Grade 1 toxicities due to prior treatment or other causes are permitted

Patient Characteristics:

* Must have ECOG Performance status of 0-2
* Must be at least 18 years of age
* Must have the following clinical laboratory values: ANC at least 1,500/mm3, platelets at least 100,000/mm3, hemoglobin at least 9 g/dL, albumin at least 3.0 g/dL, serum creatinine not more than 2.0 mg/dL, total bilirubin not more than the institutional upper limit of normal, alanine aminotransferase, aspartate aminotransferase, and alkaline phosphatase not more than 1.5 x the institutional upper limit of normal
* Must sign informed consent
* No active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease)
* No infection requiring parenteral antibiotics
* No known HIV infection or viral hepatitis
* No active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, arrhythmias requiring medication
* No known or suspected active CNS metastasis
* No pregnant or nursing female patients. Women of child-bearing potential must have negative serum or urine pregnancy test within 1 week prior to study entry. Sexually active patients (both men and women) must agree to use acceptable contraceptive methods, e.g., double barrier, during the conduct of the study
* No agent which could interfere with SN38 metabolism, including phenobarbital, valproic acid, cyclosporine or phenytoin
* No concurrent treatment for cancer or any other investigational agent for any indication within 30 days prior to receiving the first dose of study drug
* No immediate palliative treatment of any kind including surgery
* No high-dose chemotherapy regimen with stem cell support in the previous 6 months
* No abdominal or pelvic radiation therapy
* Not willing or unable to follow protocol requirements
* No known hypersensitivity to irinotecan, SN38, or liposomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-10; Primary Completion 2007-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida; Patricia LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute, Detroit, Michigan; Eric Kraut, MD, Principal Investigator — The Ohio State University, Columbus, Ohio
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - The Ohio State University, Columbus, Ohio